CLINICAL TRIAL: NCT05693714
Title: Prevelance of Adenovirus in Children With Acute Hepatitis in Assiut University Hospital
Brief Title: Adenovirus Infection in Children With Autoimmune Hepatitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rana Refaat Abdelhafeez, Assiut lecturer, Assiut University
Other Study IDs: Adenovirus infection
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2022-12

CONDITIONS: Observational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- 1: One group who have adenovirus infection
  Interventions: Diagnostic Test: Pcr

INTERVENTIONS:
Diagnostic Test: Pcr — Polymerase chain reaction
  Other Names: Pcr(polymerase chain reaction)

SUMMARY:
Adenoviruses have been linked to severe hepatitis in children. They are non-enveloped, icosahedral viruses of medium size (90-100 nm) (5). Adenoviruses usually infect the respiratory tract, eyes, urinary tract, intestines, and central nervous system (6). These diseases are

DETAILED DESCRIPTION:
Hepatitis is an inflammatory reaction of the liver that lead to a spectrum of health problems (1). Hepatitis results from a variety of causes, both infectious and non-infectious. Infectious agents include viruses and parasites. Non-infectious causes include drugs and toxic agents (2).

Viral hepatitis remains an important challenge to human health, making it a leading cause of death globally. The absolute burden of viral hepatitis is increasing gradually (3).

The most common types of viral hepatitis are hepatitis A, B, and C. The other types are hepatitis D and E, which are less frequent (2). Epstein-Barr virus (EBV) and cytomegalovirus (CMV) infections are common and are associated with liver manifestations (4).

Adenoviruses have been linked to severe hepatitis in children. They are non-enveloped, icosahedral viruses of medium size (90-100 nm) (5). Adenoviruses usually infect the respiratory tract, eyes, urinary tract, intestines, and central nervous system (6). These diseases are generally self-limiting, but severe infections can occur in immunocompromised hosts (7). Children are more susceptible to HAdVs infection because their immune systems are less developed. HAdVs cause a range of symptoms, including colds, vomiting, diarrhea, and sometimes pneumonia, but rarely hepatitis in immunocompromised patients (8) In April 2022, the WHO has reported severe acute hepatitis outbreaks among children from 11 countries across Europe and America, which have induced great public concern, HAdV is presumed to be a possible etiology of this outbreak (9).

The diagnostic methods for adenovirus include antigen detection, polymerase chain reaction (PCR), virus isolation, and serology (10).

ELIGIBILITY:
Inclusion Criteria:

- All children who are presented with symptoms suggestive of acute hepatitis like clinical jaundice, in the form of yellowish discoloration on sclera, fever, abdominal pain, diarrhea and raised liver enzymes between age group 2 years and 16 years.

Exclusion Criteria:

* -All patients under 2 years old and above 16 years.
* History of drug intake which may affect liver functions

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cross sectional study
Sampling Method: Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2023-01-20 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adenovirus infection | 2024
  Prevalence of adenovirus infection in children with autoimmune hepatitis
Adenovirus infection | 2025
  Prevalence of adenovirus infection in children with autoimmune hepatitis